CLINICAL TRIAL: NCT05583344
Title: 17 β-Hydroxysteroid Dehydrogenase Type 13 Minimization for the Treatment of NASH (HORIZON): A Double-Blind, Placebo-Controlled Phase 2b Study to Evaluate the Efficacy and Safety of GSK4532990 in Adults With Nonalcoholic Steatohepatitis
Brief Title: Phase 2b Study of GSK4532990 in Adults With NASH
Acronym: HORIZON
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 218672; 2022-002538-14 (EudraCT Number); 2023-507503-62-00 (Other: EU CT number)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Nonalcoholic Fatty Liver Disease; Non-alcoholic Fatty Liver Disease
Keywords: 17β-Hydroxysteroid Dehydrogenase type 13 Minimization for the treatment of NASH (HORIZON); GSK4532990; Non-alcoholic steatohepatitis (NASH); Non-alcoholic fatty liver disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose GSK4532990 (Experimental)
  Interventions: Drug: GSK4532990
- Low Dose GSK4532990 (Experimental)
  Interventions: Drug: GSK4532990
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK4532990 — GSK4532990 will be administered.
  Arms: High Dose GSK4532990; Low Dose GSK4532990
Drug: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure improvements in liver fibrosis and inflammation with GSK4532990 compared with placebo in participants with NASH and advanced fibrosis on biopsy (F3 or F4). The study duration will be up to 76 weeks including the screening period. The treatment duration will be up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥25 kilogram per meter square (kg/m^2) (all ethnic origins) except for Asian participants who qualify for the study with BMI ≥23 kg/m2 at Screening.
* In the opinion of the investigator, there are features of metabolic syndrome and NAFLD is the most likely cause of liver disease. Metabolic syndrome may include type 2 diabetes mellitus (T2DM), obesity, dyslipidemia and hypertension.
* A liver biopsy at baseline showing NAFLD Activity Score (NAS) >=4 with at least 1 point each in steatosis, inflammation and ballooning and either Fibrosis 3 or Fibrosis 4 using NASH CRN Scoring System.
* Able and willing to comply with all study assessments, including a liver biopsy at Week 52.

Exclusion Criteria:

* Current alcohol consumption ≥14 standard drinks (24 units, 196 g ethanol) per week for females or ≥21 standard drinks (37 units, 294g ethanol) per week for males.
* Weight reduction surgery or procedures (including gastric banding and intragastric balloon insertion) within 2 years of Screening 1 and/or planned during the study.
* History of cancer within previous 2 years from Screening 1, except basal or squamous cell carcinoma of the skin or in situ cervical carcinoma or any other type of cancer which has been treated medically or surgically with curative outcome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving ≥ 1 Stage Improvement in Histological Fibrosis with no Worsening of NASH - F3 Cohort | At Week 52
  Improvement in histological fibrosis is assessed with Clinical research network (CRN) Scoring. No worsening of NASH is defined as no increase in the NAFLD Activity Score (NAS) for steatosis, ballooning, or inflammation.
Percentage of Participants Achieving NASH Resolution with no Worsening of Fibrosis - F3 Cohort | At Week 52
  NASH resolution is defined as a ballooning score of 0 and an inflammation score of 0-1. No worsening of fibrosis is defined as no increase in CRN fibrosis score.

SECONDARY OUTCOMES:
Percentage of Participants Achieving ≥ 1 Stage Improvement in Histological Fibrosis with no Worsening of NASH - Pooled Cohort (F3 participants and F4 participants) | At Week 52
  Improvement in histological fibrosis is assessed with Clinical research network (CRN) Scoring. No worsening of NASH is defined as no increase in the NAFLD Activity Score (NAS) for steatosis, ballooning, or inflammation.
Percentage of Participants Achieving NASH Resolution with no Worsening of Fibrosis - Pooled Cohort (F3 participants and F4 participants) | At Week 52
  NASH resolution is defined as a ballooning score of 0 and an inflammation score of 0-1. No worsening of fibrosis is defined as no increase in CRN fibrosis score.
Change from baseline in Pro-peptide of type III collagen (Pro-C3) - F3 Cohort | Baseline (Day 1) and at Week 24 and 52
Change from baseline in liver fat using Magnetic resonance imaging-proton density fat fraction (MRI-PDFF) - F3 Cohort | Baseline (Day 1) and at Week 24 and 52
Change from baseline in Liver stiffness measurement (LSM) by Vibration-controlled transient elastography (VCTE) - F3 Cohort | Baseline (Day 1) and at Week 24 and 52
Change from baseline in Enhanced Liver Fibrosis (ELF) Score - F3 Cohort | Baseline (Day 1) and at Week 24 and 52
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers, including tissue inhibitor of metalloproteinases-1 (TIMP-1), type III procollagen (PIIINP), and hyaluronic acid (HA). The ELF score is used as a prognostic marker for disease progression: ELF score < 9.8 : Low risk of progression, ELF score 9.8 to < 11.3 : Moderate risk of progression and ELF score > = 11.3 : High risk of progression.
Percentage of Participants Achieving ≥30% relative reduction in liver fat from baseline using MRI-PDFF at Week 24- F3 Cohort | At Week 24
Percentage of Participants Achieving ≥30% relative reduction in liver fat from baseline using MRI-PDFF at Week 52 - F3 Cohort | At Week 52
Change from Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Gamma-glutamyl transferase (GGT) (Units Per Liter) - F3 Cohort | Baseline (Day 1) and at Week 24 and 52
Change from baseline in Pro-peptide of type III collagen (Pro-C3) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and at Week 24 and 52
Change from baseline in liver fat using Magnetic resonance imaging-proton density fat fraction (MRI-PDFF) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and at Week 24 and 52
Change from baseline in Liver stiffness measurement (LSM) by Vibration-controlled transient elastography (VCTE) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and at Week 24 and 52
Change from baseline in Enhanced Liver Fibrosis (ELF) Score - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and at Week 24 and 52
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers, including tissue inhibitor of metalloproteinases-1 (TIMP-1), type III procollagen (PIIINP), and hyaluronic acid (HA). The ELF score is used as a prognostic marker for disease progression: ELF score < 9.8 : Low risk of progression, ELF score 9.8 to < 11.3 : Moderate risk of progression and ELF score > = 11.3 : High risk of progression.
Percentage of Participants Achieving ≥30% relative reduction in liver fat from baseline using MRI-PDFF at Week 24 - Pooled Cohort (F3 participants and F4 participants) | At Week 24
Percentage of Participants Achieving ≥30% relative reduction in liver fat from baseline using MRI-PDFF at Week 52 - Pooled Cohort (F3 participants and F4 participants) | At Week 52
Change from Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Gamma-glutamyl transferase (GGT) (Units Per Liter) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and at Week 24 and 52
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) - F3 Cohort | Up to Week 66
Change from Baseline in Vital Signs - Blood Pressure (millimeters of Mercury) - F3 Cohort | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Temperature (Celsius) - F3 Cohort | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Heart Rate (Beats per minute) - F3 Cohort | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Respiratory Rate (Breaths per minute) - F3 Cohort | Baseline (Day 1) and up to Week 52
Change From Baseline in Clinical Chemistry Parameter: total bilirubin, direct Bilirubin and creatinine (Micromoles per Liter) - F3 Cohort | Baseline (Day 1) and up to Week 52
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) - F4 Cohort | Up to Week 66
Change from Baseline in Vital Signs - Blood Pressure (millimeters of Mercury) - F4 Cohort | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Temperature (Celsius) - F4 Cohort | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Heart Rate (Beats per minute) - F4 Cohort | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Respiratory Rate (Breaths per minute) - F4 Cohort | Baseline (Day 1) and up to Week 52
Change From Baseline in Clinical Chemistry Parameter: total bilirubin, direct Bilirubin and creatinine (Micromoles per Liter) - F4 Cohort | Baseline (Day 1) and up to Week 52
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) - Pooled Cohort (F3 participants and F4 participants) | Up to Week 66
Change from Baseline in Vital Signs - Blood Pressure (millimeters of Mercury) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Temperature (Celsius) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Heart Rate (Beats per minute) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and up to Week 52
Change from Baseline in Vital Signs - Respiratory Rate (Breaths per minute) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and up to Week 52
Change From Baseline in Clinical Chemistry Parameter: total bilirubin, direct Bilirubin and creatinine (Micromoles per Liter) - Pooled Cohort (F3 participants and F4 participants) | Baseline (Day 1) and up to Week 52
Area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC0-t) of GSK4532990 - F3 Cohort | Pre-dose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
Maximum observed concentration (Cmax) of GSK4532990- F3 Cohort | Pre-dose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
Percentage of Participants with Anti-drug Antibodies (ADA) to GSK4532990- F3 Cohort | Up to Week 52
Area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC0-t) of GSK4532990 - F4 Cohort | Pre-dose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
Maximum observed concentration (Cmax) of GSK4532990- F4 Cohort | Pre-dose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
Percentage of Participants with Anti-drug Antibodies (ADA) to GSK4532990- F4 Cohort | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (147):
- United States (70):
  - GSK Investigational Site, Homewood, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Rialto, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Lakewood Rch, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Bastrop, Louisiana
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Greenbelt, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, Sparta, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Springboro, Ohio
  - GSK Investigational Site, Westlake, Ohio
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Brownsville, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Edinburg, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Pilar
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (2):
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
- Canada (2):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Toronto, Ontario
- France (5):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Strasbourg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Rio Patras
  - GSK Investigational Site, Thessaloniki
- India (9):
  - GSK Investigational Site, Bhubaneswar
  - GSK Investigational Site, Chandigarh
  - GSK Investigational Site, Coimbatore
  - GSK Investigational Site, Guhawati
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Surat
- Italy (8):
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
  - GSK Investigational Site, San Giovanni Rotondo FG
- Japan (16):
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Yamanashi
- Mexico (3):
  - GSK Investigational Site, Cuernavaca Morelos
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mérida
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, San Juan, Puerto Rico
- South Korea (3):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Yongsan-Ku Seoul
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Sabadell Barcelona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Vigo
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Kocaeli
  - GSK Investigational Site, Rize
- United Kingdom (5):
  - GSK Investigational Site, Cannock
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.